CLINICAL TRIAL: NCT01263808
Title: A Randomized, Multiple-dose, Placebo- and Positive-controlled Parallel Group Study to Evaluate the Effects of Indacaterol on Cardiac Safety in Healthy Subjects
Brief Title: Cardiac Safety of Indacaterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2339
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Healthy Volunteers; Chronic Obstructive Pulmonary Disease
Keywords: Indacaterol; Moxifloxacin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Indacaterol 150 µg (Experimental): Indacaterol 150 µg
  Interventions: Drug: Indacaterol 150 µg
- Indacaterol 300 µg (Experimental): Indacaterol 300 µg
  Interventions: Drug: Indacaterol 300 µg
- Indacaterol 600 µg (Experimental): Indacaterol 600 µg
  Interventions: Drug: Indacaterol 600 µg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Placebo/moxifloxacin (Active Comparator): Placebo/moxifloxacin
  Interventions: Drug: Placebo/moxifloxacin

INTERVENTIONS:
Drug: Indacaterol 150 µg — Once daily (QD) via single-dose dry powder inhaler (SDDPI)
  Arms: Indacaterol 150 µg
Drug: Indacaterol 300 µg — QD via SDDPI
  Arms: Indacaterol 300 µg
Drug: Indacaterol 600 µg — QD via SDDPI
  Arms: Indacaterol 600 µg
Drug: Placebo — QD via SDDPI
  Arms: Placebo
Drug: Placebo/moxifloxacin — Placebo QD via SDDPI for 14 days, followed by a single dose of moxifloxacin 400 mg
  Arms: Placebo/moxifloxacin

SUMMARY:
This study compares the cardiac safety of inhaled indacaterol with that of placebo and oral moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking
* Body mass index (BMI) 18.5-32 kg/m2
* Body weight at least 50 kg

Exclusion Criteria:

* Recent/concurrent use of concomitant medications (except acetaminophen)
* Recent participation in other clinical trials
* Recent donation or loss of blood
* History/presence of a range of medical conditions, including electrocardiographic (ECG) abnormalities, diabetes mellitus, hyperthyroidism and impaired renal function

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTc interval (Fridericia's) | Change from baseline (prior to the first dose) to Day 14

SECONDARY OUTCOMES:
Change from baseline in uncorrected QT interval | Change from baseline (prior to the first dose) to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis investigative site, Miami, Florida, United States

REFERENCES:
- [Derived] Khindri S, Sabo R, Harris S, Woessner R, Jennings S, Drollmann AF. Cardiac safety of indacaterol in healthy subjects: a randomized, multidose, placebo- and positive-controlled, parallel-group thorough QT study. BMC Pulm Med. 2011 May 26;11:31. doi: 10.1186/1471-2466-11-31. PMID 21615886